CLINICAL TRIAL: NCT05108519
Title: A Prospective Study Evaluating Complications and Clinical Response in Cancer Patients Treated With Anti-VEGF-Related Therapies
Brief Title: Complications and Clinical Response in Cancer Patients Treated With Anti-VEGF-Related Therapies
Status: Recruiting | Type: Observational
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: PA18-1070; NCI-2021-06311 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2021-10-25; First posted 2021-11-05 (Actual); Last update posted 2025-08-15 (Actual); Status verified 2025-08

CONDITIONS: Hematopoietic and Lymphoid Cell Neoplasm; Malignant Solid Neoplasm
MeSH Terms: conditions — Hematologic Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Observational (medical records review): Patients' medical records are reviewed.
  Interventions: Other: Electronic Health Record Review

INTERVENTIONS:
Other: Electronic Health Record Review — Medical records are reviewed

SUMMARY:
This study collects information about complications and clinical response in cancer patients treated with anti-VEGF-related therapies. This study aims to observe side effects that may happen to patients with advanced cancer who are treated with anti-VEGF related therapy. This may help doctors learn if there are any relationships between these side effects and how the disease may respond to treatment.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To explore the incidence of clinical complications associated with anti-VEGF-related therapies in cancer patients treated at Emory University and the University of Texas M.D. Anderson Cancer Center (MDACC).

SECONDARY OBJECTIVES:

I. To explore the correlation of clinical response rates to a novel blood pressure scoring system in cancer patients treated with anti-VEGF-related therapies.

II. To explore the correlation of objective response to each toxicity grade 3 or higher in cancer patients treated with anti-VEGF-related therapies.

III. To investigate the validity of a novel multi-parameter-based blood pressure scoring system and to determine if the new scoring method is concordant with the current Common Terminology Criteria for Adverse Events (CTCAE) method.

OUTLINE:

Patients' medical records are reviewed.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be able to understand and be willing to sign a written informed consent document
* Patients must be receiving any anti-VEGF-related regimen in monotherapy or combination therapy

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients receiving any anti-VEGF-related regimen
Sampling Method: Non-Probability Sample
Enrollment: 170 (Estimated)
Dates: Start 2019-04-08 (Actual); Primary Completion 2027-02-02 (Estimated); Study Completion 2027-02-02 (Estimated)

PRIMARY OUTCOMES:
Incidence of grade 3+ adverse events (AE) at least possibly related to anti-VEGF-related treatment (overall and each type separately) | Up to 5 years
  For each toxicity, will estimate the odds ratio, associated 95% confidence interval and p-value.

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas L Palaskas, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: M D Anderson Cancer Center website — http://www.mdanderson.org